CLINICAL TRIAL: NCT00625131
Title: Nicotine Patch Pre-treatment for Smoking Cessation in PTSD
Brief Title: Nicotine Patch Pretreatment for Smoking Cessation in PTSD
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NEUA-007-07F
Record Dates: First submitted 2008-02-19; First posted 2008-02-28 (Estimated); Results first posted 2014-11-20 (Estimated); Last update posted 2014-11-20 (Estimated); Status verified 2014-11

CONDITIONS: Stress Disorders, Posttraumatic; Tobacco Use Disorder
Keywords: Stress Disorders, Posttraumatic; Tobacco Use Disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Tobacco Use Disorder | interventions — Nicotine; Cognitive Behavioral Therapy; Bupropion

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Active Nicotine Patch Group (Active Comparator): Transdermal nicotine patch
  Interventions: Drug: Nicotine; Behavioral: Cognitive Behavioral Therapy for Smoking Cessation; Drug: Bupropion Sustained Release (SR)
- Placebo Patch Group (Placebo Comparator): Transdermal placebo patch
  Interventions: Behavioral: Cognitive Behavioral Therapy for Smoking Cessation; Drug: Bupropion Sustained Release (SR); Drug: Placebo patch

INTERVENTIONS:
Drug: Nicotine — Delivered through transdermal nicotine patch
  Arms: Active Nicotine Patch Group
Behavioral: Cognitive Behavioral Therapy for Smoking Cessation — Manualized protocol for CBT in smoking cessation
  Other Names: CBT
Drug: Bupropion Sustained Release (SR) — Antidepressant
  Other Names: Zyban, Wellbutrin
Drug: Placebo patch — Pre-treatment placebo transdermal patch
  Arms: Placebo Patch Group

SUMMARY:
This study seeks to evaluate the relationship between PTSD, abstinence, and factors associated with relapse in the context of a randomized, clinical smoking cessation trial.

DETAILED DESCRIPTION:
Smokers with PTSD will be randomly assigned to 1 of 2 pre-cessation patch therapy conditions (active patch versus placebo patch) for three weeks before a target quit-smoking date. All participants to will receive bupropion beginning 1 week prior to their quit day, given that they are medically eligible to be prescribed bupropion. All participants will receive a two session brief cognitive-behavioral therapy (CBT) session and will begin standard nicotine replacement therapy (NRT) on their quit day. PTSD symptoms, mood, and smoking craving will be carefully evaluated throughout the study using electronic diary assessments on personal digital assistants (PDA). Specifically, participants will carefully monitor their symptoms, mood, craving, and use of cigarettes using electronic diaries for one week prior to the pre-cessation period, during the 3-week pre-cessation treatment period, and 6 weeks post quit date. Since no previous study has examined factors associated with smoking abstinence following treatment among PTSD smokers10, predictors of treatment response will be examined. The study is designed to address the following items:

Specific Aim 1: To evaluate whether supplemental nicotine administration (i.e., pre-cessation treatment with nicotine patch and bupropion) will result in improved quit rates among smokers with PTSD.

Hypothesis 1.1 Supplemental nicotine administration during the pre-cessation period will result in improved quit rates in the first quit week over the placebo patch condition.

Specific Aim 2: To utilize electronic diary assessment of PTSD symptoms, mood, smoking craving, and smoking during baseline, pretreatment, and quit periods to evaluate potential mechanisms of how pretreatment with the nicotine patch may increase abstinence rates.

Hypothesis 2.1 Supplemental nicotine administration will decrease craving for cigarettes during the 2 week pretreatment period as compared to the placebo patch condition.

Hypothesis 2.2 Supplemental nicotine administration will decrease the perceived improvement in mood and PTSD symptoms associated with smoking behavior, i.e., symptom relief from ad lib smoking a cigarette will be reduced during supplemental nicotine administration as compared to the placebo patch condition.

Specific Aim 3: To investigate potential predictors of smoking abstinence and relapse associated with individual differences in affective style including anxiety sensitivity, measures of distress tolerance, and self-efficacy.

Hypothesis 3.1 Increased anxiety sensitivity will be predictive of shorter abstinence from smoking.

Hypothesis 3.2 Decreased distress tolerance will be predictive of shorter abstinence.

Hypothesis 3.3 Lower self-efficacy for smoking abstinence will be predictive of shorter abstinence.

Hypothesis 3.4 Increased PTSD symptoms severity and negative affect following the quit date will be associated with shorter abstinence.

ELIGIBILITY:
Inclusion Criteria:

* Smokers who smoke 10 or more cigarettes per day in the past year;
* 18-80 years old;
* English speakers;
* medically stable;
* stable on current medication regimen

Exclusion Criteria:

* Pregnant women excluded;
* participants with organic mental disorder, schizophrenia, bipolar disorder, lifetime but not current PTSD, current substance abuse or dependence;
* medical conditions contraindicated with nicotine replacement therapy;
* use other forms of nicotine (cigars, nicotine gum, etc.)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2008-05; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jean C. Beckham, PhD, Principal Investigator — VA Medical Center, Durham
Locations (1):
- VA Medical Center, Durham, Durham, North Carolina, United States

REFERENCES:
- [Derived] Dedert EA, Dennis PA, Calhoun PS, Dennis MF, Beckham JC. A Randomized Clinical Trial of Nicotine Preloading for Smoking Cessation in People with Posttraumatic Stress Disorder. J Dual Diagn. 2018 Jul-Sep;14(3):148-157. doi: 10.1080/15504263.2018.1468947. Epub 2018 Oct 10. PMID 29693495

RESULTS

PARTICIPANT FLOW:
Groups:
- Active Nicotine Patch Group: Transdermal nicotine patch
  Nicotine: Delivered through transdermal nicotine patch
  Cognitive Behavioral Therapy for Smoking Cessation: Manualized protocol for CBT in smoking cessation
  Bupropion SR: Antidepressant
- Placebo Patch Group: Transdermal placebo patch
  Cognitive Behavioral Therapy for Smoking Cessation: Manualized protocol for CBT in smoking cessation
  Bupropion SR: Antidepressant
- Not Randomized: This arm includes patients who met screening criteria for entry into the randomization, but withdrew prior to randomization.
Period: Overall Study
Arm/Group | Active Nicotine Patch Group | Placebo Patch Group | Not Randomized
Started | 38 | 44 | 5 (These participants were not included in any analyses.)
Completed | 34 | 42 | 0
Not Completed | 4 | 2 | 5
Not completed — Lost to Follow-up | 3 | 2 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 5

BASELINE CHARACTERISTICS:
Groups:
- Arm 1: Transdermal nicotine patch
  Nicotine: Delivered through transdermal nicotine patch
  Cognitive Behavioral Therapy for Smoking Cessation: Manualized protocol for CBT in smoking cessation
  Bupropion SR: Antidepressant
- Arm 2: Transdermal placebo patch
  Cognitive Behavioral Therapy for Smoking Cessation: Manualized protocol for CBT in smoking cessation
  Bupropion SR: Antidepressant
- Total: Total of all reporting groups
Arm/Group | Arm 1 | Arm 2 | Total
Number analyzed (Participants) | 38 | 44 | 82
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.16 (9.61) | 44.48 (11.31) | 44.79 (10.51)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 21 | 38
  Male | 21 | 23 | 44
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 21 | 30 | 51
  White | 11 | 12 | 23
  More than one race | 4 | 2 | 6
  Unknown or Not Reported | 1 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2
  Not Hispanic or Latino | 35 | 44 | 79
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 38 | 44 | 82

OUTCOME MEASURES:

1. Primary Outcome: Smoking Abstinence, Self-reported
Description: Number of participants by group reporting 1 week of self-reported abstinence in the week prior to Session 12 at six weeks post-treatment
Time Frame: Week prior to Session 12 at 6 weeks post-treatment
Population: Any participants who did not attend Session 12 for any reason (i.e., lost to contact, withdrawn after beginning treatment) were counted as smoking (i.e., intent-to-treat analyses, missing = smoking).
Measure: Number; unit: participants
Arm/Group | Active Nicotine Patch Group | Placebo Patch Group
Number analyzed (Participants) | 38 | 44
participants | 5 | 11

2. Secondary Outcome: Carbon Monoxide Monitoring
Description: Number of participants whose carbon monoxide (CO) measurement indicated abstinence at Session 12 (6 weeks post-treatment)
Time Frame: Session 12 (6 weeks post-treatment)
Population: Please note that this secondary outcome (bioverification by CO reading) is not a measure of complete smoking abstinence during the study period (or during the week prior to the session - see Primary Outcome). It is independent of self-reported smoking abstinence. It is not unexpected that CO readings different than self-reported smoking.
Measure: Number; unit: participants
Arm/Group | Active Nicotine Patch Group | Placebo Patch Group
Number analyzed (Participants) | 21 | 21
participants | 8 | 5

3. Secondary Outcome: Smoking Craving
Description: Mean smoking craving score (as measured during daily ecological momentary, or diary, assessments) for participants by group during the two week period of placebo/active pre-treatment. This is the main period of interest, as it was hypothesized that use of active nicotine patch would reduce smoking cravings during the pre-quit period. The craving score is based on a single diary item "Please rate your desire to smoke right now" with a Likert scale score ranging from 1 (none) to 5 (severe). Higher craving is "worse," as lower craving is presumed to reflect decreased risk of smoking lapse or relapse.
Time Frame: Daily between visits 2-12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active Nicotine Patch Group | Placebo Patch Group
Number analyzed (Participants) | 32 | 41
units on a scale | 2.48 (1.40) | 2.59 (1.24)

ADVERSE EVENTS:
Time Frame: AE data were collected in real time during each participant session or contact from baseline to 6 month follow-up (ranging from one day to nine months). These data represent AEs reported by all participants over the entire 4 years of data collection.
Description: Serious AEs were reviewed with the PI immediately after they were reported to the study coordinator. Non-serious AEs were reviewed with the PI at weekly staff meetings.
Arm/Group | Active Nicotine Patch Group | Placebo Patch Group
Serious Adverse Events (participants affected / at risk) | 0/38 | 2/44
Other Adverse Events (participants affected / at risk) | 12/38 | 16/44
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active Nicotine Patch Group (N=38) | Placebo Patch Group (N=44)
Hospitalization for pre-existing Chronic Obstructive Pulmonary Disease (COPD) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Hospitalization for preexisting circulatory disorder (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active Nicotine Patch Group (N=38) | Placebo Patch Group (N=44)
nausea (Gastrointestinal disorders) | 0 (0) | 4 (6)
Surgical Intervention, non-study related (General disorders) | 3 (3) | 2 (2) — Several participants had minor surgical interventions during the course of the study that were not related to study participation.
Exacerbation of pre-existing PTSD symptoms (Psychiatric disorders) | 4 (4) | 7 (7)
Sleep disturbance and/or increased nightmares (Psychiatric disorders) | 7 (7) | 2 (2)
Itching and/or skin rash at site of patch placement (Skin and subcutaneous tissue disorders) | 6 (6) | 3 (3)
Orthopedic accident, not study related (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Dry mouth (Gastrointestinal disorders) | 3 (3) | 0 (0)
Gas and/or hemorrhoid pain (Gastrointestinal disorders) | 2 (4) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes